CLINICAL TRIAL: NCT04243941
Title: LCCC 1917: Dose Escalation of Low and Intermediate Risk Localized Prostate Cancer Using 68Ga-HBED-CC PSMA-PET/MRI and Stereotactic Body Radiotherapy
Brief Title: PSMA-PET/MRI Low- and Intermediate-Risk Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1917
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PMSA-PET/MRI (Experimental): Patients scheduled to receive PMSA-PET/MRI scan in addition to standard of care CT scan prior to treatment
  Interventions: Drug: 68Ga-HBED-CC-PSMA

INTERVENTIONS:
Drug: 68Ga-HBED-CC-PSMA — Radioactive tracer used during imaging to help detect PSMA expressing tumor cells
  Other Names: gallium Ga 68-labeled PSMA-11

SUMMARY:
The goal of this study is to determine the safety of using PSMA-PET/mpMRI to define radiotherapy targets, while meeting all current planning criteria. This study also intends to determine the feasibility of performing stereotactic body radiation therapy with simultaneous integrated boost on the dominant intra-prostatic lesions while meeting all current planning criteria.

DETAILED DESCRIPTION:
This study aims to determine if multi-parametric magnetic resonance imaging (mpMRI) and prostate-specific membrane antigen-positron emission tomography (PSMA-PET) imaging can help optimize the placement of the high dose inhomogeneity characterizing stereotactic body radiation therapy. All radiation plans have "hot spots" of radiation, and in current practice these regions are randomly located. This study will focus those hot spots on regions determined by mpMRI + PSMA-PET to have visible tumor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information
* Male subjects ≥ 18 years of age
* Histologically confirmed prostate adenocarcinoma
* Low or favorable intermediate risk, based on the NCCN criteria
* Subject has adequate performance status as defined by ECOG performance status of 0-2
* Subject is willing and able to comply with the protocol as determined by the Treating Investigator
* Subject speaks English (quality of life instrument is validated in English)

Exclusion Criteria:

* Contraindications for MRI
* Other prior or concomitant malignancies, with the exception of:
* non-melanoma skin cancer
* other cancer for which the subject has been disease free for ≥5 years before the first study treatment and of low potential risk for recurrence
* Inflammatory bowel disease
* Previous transurethral resection of the prostate (TURP) or surgery of the prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants only, since this is a prostate cancer study
Enrollment: 0 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Genitourinary and gastrointestinal toxicity 12 months post-treatment | Baseline to 1 year post-treatment
  Grade 2+ GU/GI late toxicity as classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 at 12 months after radiation therapy
Feasibility of meeting specified dose constraints | Baseline to 1 year post-treatment
  Proportion of subjects who meet these criteria:
  * Boost dose coverage: DIL D95% ≥ 44 Gy
  * Dose constraints:
  Urethra Dmax < 40 Gy
  Bladder Dmax < 45.6 Gy
  Bladder D10cc < 41.8 Gy
  Rectum Dmax < 38 Gy
  Rectal Mucosa D1% < 28.5 Gy
  Sigmoid Colon Dmax < 28.5 Gy

SECONDARY OUTCOMES:
Acute and late genitourinary and gastrointestinal toxicity | Baseline to 5 years post-treatment
  GU and GI toxicity as classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Will be measured during radiation therapy and at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months after radiotherapy.
Biochemical control using Prostate-Specific Antigen (PSA) levels | Baseline to 5 years post-treatment
  Biochemical control will be defined according to the Phoenix criteria at 2 and 5 years after radiation therapy
Patient-reported quality of life using the Expanded Prostate Cancer Index Composite (EPIC-26) | Baseline to 5 years post-treatment
  Measuring patient-reported quality of life using EPIC-26 prior to radiation therapy and over time in subjects with prostate cancer who have received PSMA-PET/MRI to define radiotherapy targets.
Screened Subjects | Through study completion, average of 2 years
  Measuring the proportion of screened subjects who are enrolled on the study
Patient-reported quality of life using Prostate Cancer Symptom Indices (PCSI) | Baseline to 5 years post-treatment
  Measuring patient-reported quality of life using PCSI prior to radiation therapy and over time in subjects with prostate cancer who have received PSMA-PET/MRI to define radiotherapy targets.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Repka, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials